CLINICAL TRIAL: NCT05791916
Title: Clinical, Laboratory and Echocardiographic Assessment of Biomarkers in Patients With Acute Myocardial Infarction
Brief Title: Novel Biomarkers in Patients With Acute Myocardial Infarction
Acronym: CLEAR-AMI
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 3456/20
Record Dates: First submitted 2023-03-18; First posted 2023-03-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Acute Coronary Syndrome; Biochemical Dysfunction
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Echocardiography; Myocardial Work; Biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to investigate the clinical value of novel biomarkers and echocardiographic indices, including myocardial work parameters, in patients with first acute myocardial infarction. The relationship between novel echocardiographic indices with clinical data, biochemical data in different myocardial infarction types will be attempted. Prognostic implications of those indices will be explored.

DETAILED DESCRIPTION:
This study is a prospective registry designed to evaluate and explore novel associations and prognostic tools in patients with first Acute Myocardial Infarction (AMI) with or without ST elevation, as defined by the Fourth Universal Definition of Myocardial Infarction. All eligible adult patients admitted to the Department of Cardiology at AHEPA University General Hospital of Thessaloniki with AMI will be invited to participate.

Following revascularization, a complete and comprehensive medical interview will be conducted for each patient, during which demographic characteristics, baseline medical history, medical therapy upon admission and discharge, primary aetiology, and clinical presentation of hospitalization will be recorded. Laboratory data will be collected on admission and during hospitalization, including complete blood count, biochemical control, coagulation mechanism control, hormonal control, lipid profile including Lp(a), HbA1c, N-terminal pro-B-type natriuretic peptide plasma, higher-peak value of HsTnT, IL-6, and suPAR levels on admission.

A comprehensive transthoracic echocardiographic assessment (TTE) will be performed within 24-48 hours from revascularization to evaluate the cardiac function of patients. The TTE will include 2-dimensional-speckle-tracking analysis of all cardiac chambers and non-invasive calculation of myocardial work of the left and right ventricles. The clinical value and prognostic implications of these echocardiographic indices will also be investigated during follow-up.

The primary objective is to identify novel prognostic tools by examining the association between echocardiographic indices, clinical, and biochemical data. The study aims to contribute to a better understanding of the pathophysiology of this condition and the development of effective management strategies. By comprehensively assessing the clinical, biochemical, and echocardiographic features of patients with AMI, this study will help to establish a foundation for developing targeted and effective treatments for AMI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Patients acutely admitted at the Department of Cardiology of AHEPA University General Hospital, Thessaloniki, Greece with Acute Myocardial Infarction, as those are defined by the Fourth Universal Definition of Myocardial Infarction.
3. Patients without known history of coronary artery disease

Exclusion Criteria:

1. Patients < 18 years old at time of coronary angiography
2. Patients with a previous history of coronary artery disease and/or prior revascularization
3. Inability or refusal to provide informed consent
4. Subject is pregnant and/or breastfeeding or intends to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll consecutive patients admitted to the First Department of Cardiology of AHEPA University General Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece with first Acute Myocardial Infarction with or without ST elevation, as defined by the Fourth Universal Definition of Myocardial Infarction.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Relationship between clinical, laboratory and echocardiographic biomarkers | 24 months
  Clinical, laboratory, conventional and novel echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, 2-dimensional speckle-tracking analysis of all cardiac chambers.
Relationship between clinical, laboratory, and echocardiographic biomarkers with short- and long-term prognosis of patients | 24 months
  Clinical, laboratory, and echocardiographic parameters including among others left ventricular myocardial work indices, right ventricular myocardial work indices, 2-dimensional speckle-tracking analysis of all cardiac chambers.
  Different units of measure in this outcome do not represent different outcome measures. All clinical, laboratory and echocardiographic measurements will be evaluated separately in their own unit of measurement to assess potential prognostic biomarkers in patients with acute myocardial infarction. This does not render the measurement of each parameter a different clinical outcome.

SECONDARY OUTCOMES:
All-cause mortality | 24 months
  Death by any cause
Cardiovascular mortality | 24 months
  Death directly attributed to the primary disease
Heart Failure hospitalization | 24 months
  Hospitalization due to heart failure
Acute Coronary syndrome | 24 months
  Acute Coronary Syndrome including Myocardial Infarction with or without ST elevation and Unstable Angina
MACE | 24 months
  Composite of all-cause mortality, non-fatal acute coronary syndrome and heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Ziakas, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Christos Savopoulos, MD, PhD, Study Chair — School of Medicine, Aristotle University of Thessaloniki; Vasileios Kamperidis, MD, MSc, PhD, Principal Investigator — School of Medicine, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece, Thessaloniki, Central Macedonia, Greece

REFERENCES:
- [Derived] Daios S, Anastasiou V, Moysidis DV, Didagelos M, Papazoglou AS, Stalikas N, Zegkos T, Karagiannidis E, Skoura L, Kaiafa G, Makedou K, Ziakas A, Savopoulos C, Kamperidis V. Prognostic Implications of Clinical, Laboratory and Echocardiographic Biomarkers in Patients with Acute Myocardial Infarction-Rationale and Design of the ''CLEAR-AMI Study''. J Clin Med. 2023 Sep 2;12(17):5726. doi: 10.3390/jcm12175726. PMID 37685793